CLINICAL TRIAL: NCT06537427
Title: The Crosstalk Between the Epigenome and Mitochondria as a Novel Therapeutic Target to Counteract Remote Degeneration Induced by Spinal Cord Injury
Brief Title: The Crosstalk Between the Epigenome and Mitochondria in SCI
Acronym: CEM-SCI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6884
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Injury, Spinal Cord
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group/CTRL: Healthy adults undergoing spinal anesthesia for lower limbs orthopaedic surgery.
  Interventions: Other: Data collection
- Patients with an acute spinal cord injury/SCI: Patients with an acute, traumatic SCI
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The data to be collected are the following:
  * Demographic data: gender and age of the patient at diagnosis of SCI;
  * Drug assumption and drug abuse at the time of SCI;
  * A complete assessment of patients' comorbidities;
  * Complete neurological examination on admission and at 6-8 months follow-up according to ASIA protocol;
  * Neuro-radiological data: spinal CT and MRI performed within 48 hours of admission to document the type, level and extent of the lesion of the spine and the spinal cord;
  * CSF pressure, chemical and biological markers;
  * Serum chemical and biological markers;
  * Data coming from surgical procedure: type of decompression, type of stabilization, extension of the stabilization, surgical approach, staged surgery, timing of surgery, length of surgery, eventual intraoperative, postoperative or long-term surgical-related complications [13];
  * Data on hospitalization: length of stay, hospital-acquired infections, any adverse event occurred during hospitalisation.

SUMMARY:
SCI is a devastating neurological disorder for which there are not yet restorative therapies. Thus, there is a need to explore new therapeutic strategies to treat SCI patients. To this end an appropriate selection and enrolment of suitable participants is crucial for the success of the therapeutic protocol. The selection of participants in SCI trials is often based on injury categories (e.g. sensorimotor complete vs incomplete), and neglects biological aspects (e.g. biomarkers released into the CSF and/or blood) that may be amenable to specific therapeutic interventions. On a biomolecular standpoint, it is renown that CNS lacks the ability to sustain a complete regenerative response after damage, which is partially due to the inability of damaged neurons to sustain an epigenetic pro-regenerative response.

The background of the present protocol study stands in pre-existing data which showed a crosstalk between the epigenome gene and mitochondria activated upon SCI. The clinical branch of this study protocol aims to investigate if and how targeted proteomic changes following the acute and chronic phase of SCI may play a role in determining the severity of neurologic impairments, as determined with ASIA gradingscale system, at the time of patients' presentation and in the conversion of ASIA grade during follow-up. A previous pilot study conducted by Wichmann et al. has shed light on proteomics after SCI enabling a profiling of inflammatory responses after spinal cord injury, timing of proteomics changes involved in inflammatory responses and differences between proteins title in CSF and peripheral blood. On the other hand, authors failed to prove a correlation between inflammatory proteins expression and timing of expression and neurologic status. However, previous studies proved that proteome expression variations SCI-induced can be detected into patients' CSF and serum and that biomarkers released into the CSF and/or blood may provide a plethora of information as to the patients' biological response to SCI. These samples may contain a unique fingerprint that can be used by scientists and clinicians to elucidate the mechanisms underlying irreversible central nervous system (CNS) degeneration following SCI. This could allow treatments to target specific molecules which promote CNS degeneration. Within this context the identification of prognostic biomarkers of SCI will help to assign SCI patients to the correct therapeutic treatment that, in association with canonical therapies, may synergistically act to improve functional recovery.

The aim of the present study is to investigate the presence of prognostic markers in SCI patient-derived serum and CSF with respect to a control group of healthy patients.

DETAILED DESCRIPTION:
SCI is a devastating neurological disorder for which there are not yet restorative therapies. Thus, there is a need to explore new therapeutic strategies to treat SCI patients. To this end an appropriate selection and enrolment of suitable participants is crucial for the success of the therapeutic protocol [1,2]. The selection of participants in SCI trials is often based on injury categories (e.g. sensorimotor complete vs incomplete), and neglects biological aspects (e.g. biomarkers released into the CSF and/or blood) that may be amenable to specific therapeutic interventions. On a biomolecular standpoint, it is renown that CNS lacks the ability to sustain a complete regenerative response after damage, which is partially due to the inability of damaged neurons to sustain an epigenetic pro-regenerative response [3].

The background of the present protocol study stands in pre-existing data which showed a crosstalk between the epigenome gene and mitochondria activated upon SCI. In particular, previous experimental studies conducted on mice red nuclei (RN) demonstrated proteome changes at 7 days and 28 days post-SCI. Further pathway analysis pointed out to the epigenetic enzyme KDM5A as the upstream regulator of this phenotype. KDM5A is a H3K4me3 demethylase protein that plays a fundamental role in mitochondria biogenesis and function whose activity is regulated by mitochondrial metabolites [4,5]. Thereby, preliminary data suggest that downregulation of KDM5A activity and increased mitochondrial metabolism are involved in early neuronal response to remote damage. However, its role in brain pathologies such as in SCI remains still unexplored. Since it is well-established that structural and functional damages of mitochondria is an early event that contributed to neuronal cell death, hindering the possibility of axonal regeneration [6], the molecular background of the experimental branch of the present protocol study stands in the investigation of epigenetic regulation by KDM5A and mitochondrial function. The clinical branch of this study protocol aims to investigate if and how targeted proteomic changes following the acute and chronic phase of SCI may play a role in determining the severity of neurologic impairments, as determined with ASIA grading scale system, at the time of patients' presentation and in the conversion of ASIA grade during follow-up. A previous pilot study conducted by Wichmann et al. has shed light on proteomics after SCI enabling a profiling of inflammatory responses after spinal cord injury, timing of proteomics changes involved in inflammatory responses and differences between proteins title in CSF and peripheral blood. On the other hand, authors failed to prove a correlation between inflammatory proteins expression and timing of expression and neurologic status [7]. However, their paper proved that proteome expression variations SCI-induced can be detected into patients' CSF and serum and that biomarkers released into the CSF and/or blood may provide a plethora of information as to the patients' biological response to SCI. These samples may contain a unique fingerprint that can be used by scientists and clinicians to elucidate the mechanisms underlying irreversible central nervous system (CNS) degeneration following SCI. This could allow treatments to target specific molecules which promote CNS degeneration. Within this context the identification of prognostic biomarkers of SCI will help to assign SCI patients to the correct therapeutic treatment that, in association with canonical therapies, may synergistically act to improve functional recovery.

The aim of the present study is to investigate the presence of prognostic markers in SCI patient-derived serum and CSF with respect to a control group of healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* ASIA impairment scale grade A, B, or C upon admission;
* neurological level of injury between C1-L1;
* patient older than 18 years;
* ability to collect a valid, reliable baseline neurologic examination within 24h of injury.

Exclusion Criteria:

* Concomitant TBI;
* major axial or appendicular trauma;
* in case of sedation or intoxication making unreliable the neurological examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SCI patients will receive at admission an intrathecal lumbar drain below L2, that will remain in place for 5 days. Intensive care clinical setting will allow MAP continuous monitoring, whose augmentation above 85 mmHg is a well-established standard of care in SCI patients. CSF drainage will be employed for 5 days maintaining intrathecal pressure at a mean value of 5.3 mmHg with respect to the CTRL group in which the intrathecal pressure had a mean value of 15 mmHg .Lumbar intrathecal insertion will have the dual clinical objective of 1) monitoring CSFP for evaluation of SCPP and 2) collecting CSF samples if needed in order to reduce CSFP and to keep SCPP above 85 mmHg. 3 ml of blood serum will be collected daily for exams.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the proteome profile in serum and CSF samples of SCI patients | Months 1-24
  To evaluate molecular variations in CSF and/or serum SCI-derived patients, both in acute and chronic phase after injury, patients with acute SCI will be enrolled and they will be followed until the chronic stage. CSF and serum biomarkers of SCI-group will be compared to those of the control group (non-SCI group) undergoing spinal anesthesia for lower limbs orthopedic surgery, in which few milliliters of CSF and serum will be collected.

SECONDARY OUTCOMES:
Correlation of the proteome profile of SCI patient's with their clinical profile. | Months 1-24
  Once identified key biomarkers in the CSF and/or the serum of SCI patients, data on proteome profile will be combined with clinical data. This correlation will allow to gain new insights into molecular aspects of the disease and ultimately to draw a complete overview of each single patient for designing personalized treatments.
  - Comparative proteomic and metabolic analysis of data on mice samples with data on patients' samples. This analysis aims at addressing specific elements of the translational response which could represent novel prognostic biomarkers in future experimental studies.

IPD SHARING:
Plan to Share IPD: Undecided